CLINICAL TRIAL: NCT02929407
Title: A Placebo Controlled, Double-blind, Randomised Trial Investigating Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics After Intravenous Administration of FE 204205 in Patients With Cirrhotic Portal Hypertension
Brief Title: A Study to Investigate the Safety and Effect of the Study Drug (FE 204205) in Patients With Cirrhotic Portal Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial terminated due to difficult recruitment
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000249; 2016-001078-13 (EudraCT Number)
Record Dates: First submitted 2016-09-13; First posted 2016-10-11 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-06

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FE 204205 (Experimental)
  Interventions: Drug: FE 204205
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FE 204205 — In Part 1 of the trial, each subject will receive increasing IV doses of FE 204205, given once daily as 2 hour infusion, on three consecutive days.
  In Part 2 of the trial, each subject will receive a 2 hour IV infusion of the maximum tolerated dose of FE 204205 as defined in Part 1 of the trial.
  Arms: FE 204205
Drug: Placebo — In Part 2 of the trial, each subject will receive a 2 hour IV infusion of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate safety, tolerability, pharmacodynamics (PD), and pharmacokinetics (PK) after intravenous (IV) administration of FE 204205 in patients with cirrhotic portal hypertension.

DETAILED DESCRIPTION:
The trial aimed to evaluate the safety, tolerability, PK and PD of IV FE 204205 in cirrhotic patients with portal hypertension and was planned in 2 parts:

Part 1 of the trial was open-label where six subjects were planned to receive three ascending doses of FE 204205, given as infusion over 2 hours on three consecutive days.

Part 2 was planned as a randomised, placebo-controlled, double-blind investigation evaluating the effects of a single dose of FE 204205 on portal haemodynamics in 20 subjects who would have received either the maximum tolerated dose (as defined in Part 1) of FE 204205 (n=16) or placebo (n=4).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed evidence of cirrhosis
* From medical history anticipated hepatic venous pressure gradient greater than equal to (≥)12 mmHg

Exclusion Criteria:

* Co-existing disease e.g. significant organ failure and decompensated cirrhosis
* Type 1 hepatorenal syndrome
* Acute-on-chronic liver failure
* Hepatic encephalopathy ≥grade 2
* Hepatocellular carcinoma
* History of underlying chronic heart disease
* Use of vasopressin or terlipressin within 7 days prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hospital Clinic de Barcelona, Departamento hepatología, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was terminated early due to low recruitment. Only four subjects were enrolled into the open-label, exploratory Part 1 of the trial (all receiving different dosing regimens), and no subjects were enrolled into the randomized, double-blind, placebo-controlled Part 2 of the trial prior to early termination.
Pre-assignment Details: A total of five subjects were screened, of which, four subjects were enrolled in Part 1 of the trial.
Groups:
- FE 204205: FE 204205, given once daily as 2 hour intravenous (IV) infusion, on three consecutive days. The dose in each subject was escalated from one day to the next if all dose escalation criteria were met.
  The dosing regimen for each subject is given below:
  Subject 101: Day 1: 0.0325 mg; Subject 102: Day 1: 0.01 mg, Day 2: 0.026 mg, Day 3: 0.05 mg; Subject 103: Day 1: 0.01 mg, Day 2: 0.01 mg, Day 3: 0.01 mg; Subject 105: Day 1: 0.01 mg, Day 2: 0.01 mg, Day 3: 0.026 mg.
Period: Overall Study
Arm/Group | FE 204205
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- FE 204205: FE 204205, given once daily as 2 hour IV infusion, on three consecutive days. The dose in each subject was escalated from one day to the next if all dose escalation criteria were met.
  The dosing regimen for each subject is given below:
  Subject 101: Day 1: 0.0325 mg; Subject 102: Day 1: 0.01 mg, Day 2: 0.026 mg, Day 3: 0.05 mg; Subject 103: Day 1: 0.01 mg, Day 2: 0.01 mg, Day 3: 0.01 mg; Subject 105: Day 1: 0.01 mg, Day 2: 0.01 mg, Day 3: 0.026 mg.
Arm/Group | FE 204205
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Venous Pressure Gradient (HVPG)
Description: The trial was terminated early due to low recruitment. Only four subjects were enrolled into the open-label, exploratory Part 1 of the trial, and only three of these four subjects (all receiving different dosing regimens) completed the trial and the HVPG assessments prior to the early termination decision. No subjects were enrolled into the randomized, double-blind, placebo-controlled Part 2 of the trial. As only Part 2 of the trial would have been appropriately powered, and the three subjects with HVPG assessments from Part 1 all received different dosing regimens, no meaningful statistical analysis could be conducted.
Time Frame: From baseline (pre-dose) to 2 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

2. Primary Outcome: Type, Frequency and Intensity of Adverse Events (AEs)
Description: The trial was terminated early due to low recruitment. Only four subjects (all received different dosing regimens) were enrolled into open-label, exploratory Part 1 of the trial, prior to the early termination. No subjects were enrolled in the randomized, double-blind, placebo-controlled Part 2 of the trial. Thus no meaningful statistical analysis could be conducted.
  Due to the low number of subjects and individual dosing regimens, AEs were pooled for all dose levels.
Time Frame: Up to Day 14
Population: There were too few subjects for statistical analysis (see measure description).
Measure: Count of Participants; unit: Participants
Arm/Group | FE 204205
Number analyzed (Participants) | 4
Participants
  Frequency of AEs | 3
  Intensity of AEs (Mild) | 1
  Intensity of AEs (Moderate) | 1
  Intensity of AEs (Severe) | 1
  Type of AEs (Serious) | 2
  Type of AEs (Non-serious) | 2

3. Primary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: The trial was terminated early due to low recruitment. Only four subjects (all received different dosing regimens) were enrolled into open-label, exploratory Part 1 of the trial, prior to the early termination. No subjects were enrolled in the randomized, double-blind, placebo-controlled Part 2 of the trial. Thus no meaningful statistical analysis could be conducted.
Time Frame: From baseline (pre-dose) up to Day 14
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Plasma Lactate Levels
Description: as for outcome 3
Time Frame: From baseline (pre-dose) to 3 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

5. Primary Outcome: Pharmacokinetics: Maximum Concentration Observed (Cmax)
Description: The trial was terminated early due to low recruitment. Only four subjects (all received different dosing regimens) were enrolled into open-label, exploratory Part 1 of the trial, prior to the early termination. No subjets were enrolled in the randomized, double-blind, placebo-controlled Part 2 of the trial. Thus no meaningful statistical analysis could be conducted.
Time Frame: Pre-dose, 0.5, 1, 2, 3, and 4 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

6. Primary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve to Infinity (AUC)
Description: The trial was terminated early due to low recruitment. Only four subjects were enrolled (all received different dosing regimens) into open-label, exploratory Part 1 of the trial, prior to the early termination. No subjects were enrolled in the randomized, double-blind, placebo-controlled Part 2 of the trial. Thus no meaningful statistical analysis could be conducted.
Time Frame: Pre-dose, 0.5, 1, 2, 3, and 4 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

7. Primary Outcome: Pharmacokinetics: Total Systemic Clearance (CL)
Description: as for outcome 3
Time Frame: Pre-dose, 0.5, 1, 2, 3, and 4 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

8. Primary Outcome: Pharmacokinetics: Elimination Half-life (t1/2)
Description: as for outcome 6
Time Frame: Pre-dose, 0.5, 1, 2, 3, and 4 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

9. Primary Outcome: Pharmacokinetics: Volume of Distribution Associated With the Terminal Phase (Vz)
Description: as for outcome 6
Time Frame: Pre-dose, 0.5, 1, 2, 3, and 4 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

10. Primary Outcome: Change in Electrocardiogram (ECG) Parameters
Description: as for outcome 6
Time Frame: From baseline (pre-dose) up to Day 14
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

11. Primary Outcome: Change in Blood Gas (PaO2)
Description: as for outcome 6
Time Frame: From baseline (pre-dose) to 3 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

12. Primary Outcome: Change in Blood Gas (PaCO2)
Description: as for outcome 3
Time Frame: From baseline (pre-dose) to 3 hours after start of infusion
Population: There were too few subjects for statistical analysis (see measure description).
Arm/Group | FE 204205
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were recorded from obtaining the informed consent to the follow-up visit. In part 1 of the trial, AEs were recorded from obtaining the informed consent (up to 21 days before first administration of FE 204205) to the end-of-trial visit (between 7 and 14 days after first administration of FE 204205). Part 2 of the trial was never initiated.
Description: An AE was defined as any untoward medical occurrence in a subject participating in a clinical trial. An AE could be any unfavourable and unintended sign, symptom or disease temporally associated with the use of the investigational medicinal product (IMP), whether or not considered to be caused by the IMP.
  Due to the low number of subjects and individual dosing regimens, AEs were pooled for all dose levels.
Arm/Group | FE 204205
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 204205 (N=4)
Arterial Hypertension (Vascular disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 204205 (N=4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Asterixis (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT02929407/Prot_SAP_000.pdf